CLINICAL TRIAL: NCT05783544
Title: Role of A. Lumbricoides in the Development of Pulmonary Aspergillosis in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Impact of A. Lumbricoides on Pulmonary Aspergillosis Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Responsible Party: Principal Investigator, Svetlana Osipova, MD, PhD, DS, Head of Department of Immunology of Parasitic and Fungal Diseases, Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01032023
Record Dates: First submitted 2023-03-01; First posted 2023-03-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: COPD Exacerbation Acute; Ascaris Lumbricoides Infection; Chronic Pulmonary Aspergillosis
Keywords: COPD; aspergillosis; ascariasis; cytokines; helminths
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Aspergillosis; Ascariasis | interventions — Interferon-gamma Release Tests

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- COPD patients without any comorbidities (Active Comparator)
  Interventions: Diagnostic Test: Interleukin-1B; Diagnostic Test: Interleukin-4; Diagnostic Test: Interleukin-6; Diagnostic Test: tumor necrosis factor - a; Diagnostic Test: interferon- gamma
- COPD patients with chronic pulmonary aspergillosis (Active Comparator)
  Interventions: Diagnostic Test: Interleukin-1B; Diagnostic Test: Interleukin-4; Diagnostic Test: Interleukin-6; Diagnostic Test: tumor necrosis factor - a; Diagnostic Test: interferon- gamma
- COPD patients with ascariasis (Active Comparator)
  Interventions: Diagnostic Test: Interleukin-1B; Diagnostic Test: Interleukin-4; Diagnostic Test: Interleukin-6; Diagnostic Test: tumor necrosis factor - a; Diagnostic Test: interferon- gamma
- COPD patients with chronic pulmonary aspergillosis and ascariasis (Active Comparator)
  Interventions: Diagnostic Test: Interleukin-1B; Diagnostic Test: Interleukin-4; Diagnostic Test: Interleukin-6; Diagnostic Test: tumor necrosis factor - a; Diagnostic Test: interferon- gamma
- healthy control (Active Comparator)
  Interventions: Diagnostic Test: Interleukin-1B; Diagnostic Test: Interleukin-4; Diagnostic Test: Interleukin-6; Diagnostic Test: tumor necrosis factor - a; Diagnostic Test: interferon- gamma

INTERVENTIONS:
Diagnostic Test: Interleukin-1B — Level of serum interleukin-1B will be detected
Diagnostic Test: Interleukin-4 — Level of serum interleukin-4 will be detected
Diagnostic Test: Interleukin-6 — Level of serum interleukin-4 will be detected
Diagnostic Test: tumor necrosis factor - a — Level of serum tumor necrosis factor - a will be detected
Diagnostic Test: interferon- gamma — Level of serum interferon- gamma will be detected

SUMMARY:
The prevalence of ascariasis in COPD patients with and without concomitant pulmonary aspergillosis and in controls will be determined. To assess the influence of ascaridosis on the development of pulmonary aspergillosis in COPD patients cytokine status of patients will be studied.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* COPD patients with aspergillosis
* COPD patients with ascariasis
* COPD patients with mix-infection
* Healthy individuals (controls)

Exclusion Criteria:

* COPD patients with other autoimmune diseases
* COPD patients with oncological diseases
* COPD patients with other co-infections

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum interleukin-1B levels in COPD patients and controls | up to 12 months
  Serum interleukin-1B (pg/mL) levels will be measured in COPD patients without concomitant infection, COPD patients with pulmonary aspergillosis, COPD patients with ascariasis, COPD patients with ascariasis and pulmonary aspergillosis, and healthy individuals.
Serum interleukin-4 levels in COPD patients and controls | up to 12 months
  Serum interleukin-4 (pg/mL) levels will be measured in COPD patients without concomitant infection, COPD patients with pulmonary aspergillosis, COPD patients with ascariasis, COPD patients with ascariasis and pulmonary aspergillosis, and healthy individuals.
Serum interleukin-6 levels in COPD patients and controls | up to 12 months
  Serum interleukin-6 (pg/mL) levels will be measured in COPD patients without concomitant infection, COPD patients with pulmonary aspergillosis, COPD patients with ascariasis, COPD patients with ascariasis and pulmonary aspergillosis, and healthy individuals.
Serum tumor necrosis factor-a levels in COPD patients and controls | up to 12 months
  Serum tumor necrosis factor-a (pg/mL) levels will be measured in COPD patients without concomitant infection, COPD patients with pulmonary aspergillosis, COPD patients with ascariasis, COPD patients with ascariasis and pulmonary aspergillosis, and healthy individuals.
Serum interferon-gamma levels in COPD patients and controls | up to 12 months
  Serum interferon-gamma (pg/mL) levels will be measured in COPD patients without concomitant infection, COPD patients with pulmonary aspergillosis, COPD patients with ascariasis, COPD patients with ascariasis and pulmonary aspergillosis, and healthy individuals.
Correlation between cytokine status with chronic pulmonary aspergilosis insidence rate in COPD patients with and without ascariasis | up to 12 months
  The correlation between serum interleukin-1B, interleukin-4, interleukin-6, tumor necrosis factor-a and interferon-y levels with chronic pulmonary aspergilosis insidence rate in COPD patients with and without ascariasis will be assessed.

SECONDARY OUTCOMES:
Rate of ascariasis infestation among COPD patients and controls | up to 12 months
  The frequency of ascariasis infestation among COPD patients with and without pulmonary aspergillosis, as well as healthy individuals, will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research institute of epidemiology, microbiology and infectious diseases, Tashkent, Uchtepa, Uzbekistan

IPD SHARING:
Plan to Share IPD: No